CLINICAL TRIAL: NCT05878301
Title: Postprandial Glucose, Insulin Response to Meal Sequence Among Healthy UAE Adults: A Randomized Controlled Crossover Trial
Brief Title: Postprandial Glucose, Insulin Response to Meal Sequence Among Healthy UAE Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sharjah (Other)
Responsible Party: Principal Investigator, Ayah Shaheen, clinical dietitian, University of Sharjah
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: REC-22-10-18-S
Record Dates: First submitted 2023-05-17; First posted 2023-05-26 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Postprandial Hyperglycemia
MeSH Terms: conditions — Hyperglycemia | interventions — Vegetables

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- standard mixed meal (SMM) (Other): standard mixed meal (SMM) consumed within 15 min to compared to the vegetable protein first followed 10 min later by carbohydrates it with the effect on postprandial glucose ,insulin and hunger rating
  Interventions: Other: vegetable and protein first followed by carbohydrates (VPF) meal sequence

INTERVENTIONS:
Other: vegetable and protein first followed by carbohydrates (VPF) meal sequence — vegetable and protein first followed10 min later by carbohydrates (VPF) meal sequence
  Other Names: VPF

SUMMARY:
the goal of this Randomized controlled cross over trial is to compare the effects of meal sequences VPF meal vs. SMM on the incremental area under the curve of postprandial glucose response among healthy adults in the UAE. the main question it aims to answer is what is the effect of meal sequence of vegetable and protein first followed by carbohydrates (VPF) compared to a standard mixed meal (SMM) on the postprandial glucose level and insulin response among healthy adults in the UAE. Participants will consume two is caloric test meals in random order (SMM and VPF meal sequences) separated by a 7-10-day washout period then blood sample will be collected at fasting ,30min,60min and 120mon for glucose and insulin and hunger ration will be done as well .Researchers will compare the effect of the two meals on postprandial blood glucose, insuline and hunger rating.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were age of 18-59 years
* Emirati, Gulf Cooperation Council (GCC), and Arabs ethnicity
* BMI: 18.5-29.9 kg/m2
* Fasting blood glucose level less than 100 mg/dL
* Non-smoker
* no genetic or metabolic diseases
* no known medical condition.

Exclusion Criteria:

* any participants with pre-existing diabetes
* Pregnant and breastfeeding women
* Participants with behaviors or/and health conditions that are known to affect glucose or -- insulin concentrations, such as smoking, gastrointestinal conditions, bariatric surgery, gastroparesis and reactive hypoglycemia
* Participants who consumed medication that might affect glucose or insulin response
* Participants with reported allergy or intolerance to any of the meal components (White Basmati rice, grilled chicken, cucumber, tomato, and lettuce salad with lemon olive oil dressing).

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
To compare the effects of meal sequences VPF meal vs. SMM on the incremental area under the curve of postprandial glucose response among healthy adults in the UAE. | 7-10 days
  incremental area under the curve

SECONDARY OUTCOMES:
To compare the effects of the VPF meal sequence vs. SMM sequence on the incremental area under the curve of postprandial insulin response. | 2 month
  incremental area under the curve
To compare the postprandial hunger response of the VPF meal sequence vs SMM sequence on the area under the curve using a validated visual analog scale for hunger and fullness (VAS) | 7-10 days
  ]area under the curve

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetes center ,university of sharjah, Sharjah city, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shukla AP, Andono J, Touhamy SH, Casper A, Iliescu RG, Mauer E, Shan Zhu Y, Ludwig DS, Aronne LJ. Carbohydrate-last meal pattern lowers postprandial glucose and insulin excursions in type 2 diabetes. BMJ Open Diabetes Res Care. 2017 Sep 14;5(1):e000440. doi: 10.1136/bmjdrc-2017-000440. eCollection 2017. PMID 28989726